CLINICAL TRIAL: NCT02383706
Title: Obstructive Sleep Apnea in Pregnancy: Development of a Pregnancy-Specific Screening Tool
Brief Title: Obstructive Sleep Apnea in Pregnancy
Acronym: OSAinPreg
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00056786
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-03

CONDITIONS: Sleep Apnea, Obstructive; Pregnancy; Obesity, Morbid
Keywords: Sleep Apnea, Obstructive; Pregnancy; Obesity, Morbid; Complications, pregnancy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity, Morbid; Pregnancy Complications | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects: Pregnant women, BMI greater than or equal to 40 undergo questionnaires, physical exam, and ApneaLink Air, at home, overnight polysomnography study.
  Interventions: Device: ApneaLink Air; Behavioral: Berlin Quesionnaire; Behavioral: Epworth Sleepiness Scale; Behavioral: STOP-BANG questionnaire; Other: Physical exam

INTERVENTIONS:
Device: ApneaLink Air — Overnight, home polysomnography device
Behavioral: Berlin Quesionnaire — OSA screening questionnaire
Behavioral: Epworth Sleepiness Scale — OSA screening questionnaire
Behavioral: STOP-BANG questionnaire — OSA screening questionnaire
Other: Physical exam — Physical exam of neck, mouth and upper airway

SUMMARY:
Obstructive sleep apnea (OSA) is a risk factor for complications during pregnancy and current screening tools for OSA have not been shown to be reliable in pregnant women. The primary aim of this study is to develop a valid screening tool to identify at-risk pregnant women, so that they can be further evaluated and treated. Women with OSA may also be at risk for respiratory complications related to opiate administration for post-cesarean delivery pain. A secondary aim of this study is to evaluate post-operative minute ventilation in women who undergo cesarean delivery using a novel method of non-invasive minute ventilation monitoring.

DETAILED DESCRIPTION:
Following recruitment and informed consent, subjects will complete 3 screening questionnaires for OSA: the Berlin and STOP-BANG questionnaires, and the Epworth Sleepiness Scale. They will also undergo a physical exam by one of the study investigators including examination of the neck and upper airway to assess neck circumference, retrognathia, thyromental space, tongue scalloping, MMS, modified MMS, tonsil size and lateral pharyngeal wall narrowing.

Subjects will all receive ApneaLink™ Air (ResMed, Poway, CA), a FDA-approved, non-invasive, portable, home polysomnography device, and instructions for using the device during one night of sleep. They will be given contact information if they have questions regarding use of the device. Subjects will receive a prepaid FedEx envelope to return the device. They will receive a parking voucher worth up to a maximum of $7 during this appointment. Subjects will be compensated ($50 check by mail) once the device is received. A follow-up phone call will be made by the PI to inform the subject of the results of the home polysomnography study. Subjects who screen positive (AHI > 5) by home polysomnography will be referred to Duke Sleep Medicine for further evaluation. Pregnancy outcomes will be followed for all subjects.

Enrolled subjects who go on to have a cesarean delivery will be studied using ExSpiron (Respiratory Motion, Inc., Waltham, MA), a FDA-approved, non-invasive respiratory volume monitor for 24 hours. The monitor has three adhesive pads that attach to the chest wall and a cord that attaches to the monitoring device, similar to an electrocardiogram. The monitor can be detached and the study suspended when patients ambulate to the restroom, and should not interfere with breastfeeding. The monitor will be connected to the patient in the pre-operative holding area, and the monitor will be calibrated with baseline spirometry measurements using a Wright spirometer over one minute. The subject will wear the device for the duration of the surgery, in the recovery room, and for 24 following surgery. The non-invasive respiratory volume monitor will be collected by study personnel at the conclusion of the 24 hours, and no data collected from the monitor will be used for clinical decision-making. Standard of care will be followed for the antepartum, intrapartum and postpartum management of those patients. Patients will continue to be monitored using the investigators' standard protocol for patients who have received neuraxial morphine which consists of continuous monitoring for 2 hours, followed by monitoring every 2 hours for 24 hours of the following: vital signs, oxygen saturation, respiratory rate, pain score and sedation score. The investigators also have nursing standing orders for naloxone administration for respiratory rate < 8 breaths/min or Richmond Agitation Sedation Scale (RASS) ≤ -3, together with immediate notification of medical staff, as well an order to notify medical staff for oxygen saturation < 90% or RASS < -2.

ELIGIBILITY:
Inclusion Criteria:

* gestational age 24 to 35 weeks
* BMI > or equal to 40 kg/m2
* 18 years or older

Exclusion Criteria:

* Non-English speaking subjects
* Established diagnosis of OSA
* chronic narcotic use

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women, ages 18-50 years old, BMI > or equal to 40 kg/m2, without a prior diagnosis of obstructive sleep apnea or chronic narcotic use.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dominguez JE, Grotegut CA, Cooter M, Krystal AD, Habib AS. Screening extremely obese pregnant women for obstructive sleep apnea. Am J Obstet Gynecol. 2018 Dec;219(6):613.e1-613.e10. doi: 10.1016/j.ajog.2018.09.001. Epub 2018 Sep 11. PMID 30217579

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects
Started | 108
Completed | 80
Not Completed | 28

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Arm/Group | Subjects
Number analyzed (Participants) | 80
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Reported separately for participants with Obstructive Sleep Apnea and those without.
  years
    No Obstructive Sleep Apnea: number analyzed (Participants) | 61
    No Obstructive Sleep Apnea | 27 [26 to 32]
    Obstructive Sleep Apnea: number analyzed (Participants) | 19
    Obstructive Sleep Apnea | 33 [29 to 35]
    All subjects | 29.5 [24 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 78
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 52
  White | 20
  More than one race | 4
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80
Pre-pregnancy Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] — Population: Reported separately for participants with Obstructive Sleep Apnea and those without.
  kg/m^2
    Obstructive Sleep Apnea: number analyzed (Participants) | 19
    Obstructive Sleep Apnea | 53 [45 to 55]
    No Obstructive Sleep Apnea: number analyzed (Participants) | 61
    No Obstructive Sleep Apnea | 45 [41 to 51]
    All subjects | 46 [42 to 52]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Negative Obstructive Sleep Apnea (OSA) Home Sleep Test Result
Description: Determined using the Apnea-Hypopnea Index (AHI). Participants were considered OSA-negative if experienced less than five events per hour.
Time Frame: Women studied at one time point between 24 weeks and 35 weeks gestation.
Measure: Count of Participants; unit: Participants
Groups:
- Subjects: Pregnant women, BMI greater than or equal to 40 undergo questionnaires, physical exam, and ApneaLink Air, at home, overnight polysomnography study.
  ApneaLink Air: Overnight, home polysomnography device Berlin Quesionnaire: OSA screening questionnaire Epworth Sleepiness Scale: OSA screening questionnaire STOP-BANG questionnaire: OSA screening questionnaire Physical exam: Physical exam of neck, mouth and upper airway
Arm/Group | Subjects
Number analyzed (Participants) | 80
Participants | 61

2. Primary Outcome: Number of Participants With a Positive Obstructive Sleep Apnea (OSA) Home Sleep Test Result
Description: Determined using the Apnea-Hypopnea Index (AHI). Participants were considered OSA-positive if experienced five or more events per hour.
Time Frame: Women studied at one time point between 24 weeks and 35 weeks gestation.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects
Number analyzed (Participants) | 80
Participants | 19

3. Secondary Outcome: Post-op Minute Ventilation Following C-section
Description: To evaluate post-operative minute ventilation in women who undergo cesarean delivery using a novel method of non-invasive minute ventilation monitoring
Time Frame: Women studied for 24-hours following their cesarean delivery.
Population: Data not collected
Arm/Group | Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From time of enrollment until delivery, no longer than 6 months
Arm/Group | Subjects
All-Cause Mortality (participants affected / at risk) | 0/108
Serious Adverse Events (participants affected / at risk) | 0/108
Other Adverse Events (participants affected / at risk) | 0/108

LIMITATIONS AND CAVEATS:
80 subjects Home sleep testing used Low acceptance of home sleep test by subjects (28 subjects did not wear device more than 2 hours) One time point in pregnancy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT02383706/Prot_SAP_000.pdf